CLINICAL TRIAL: NCT02582177
Title: Phase 3 Study, Randomized, Double-blind, Parallel to Evaluate Ketoconazole and Betamethasone Dipropionate(Candicort®) Compared to Clotrimazole and Dexamethasone Acetate(Baycuten N®) in Relief of Fungal Infections/Dermatophytosis Symptoms.
Brief Title: Effectiveness Study of Ketoconazole and Betamethasone to Treat Fungal Infection and Dermatophytosis
Acronym: DaVinci
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACH-CND-03(05/15)
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Tinea
Keywords: Fungal infection; Skin infection; Dermatophytoses
MeSH Terms: conditions — Tinea; Mycoses; Cellulitis | interventions — Ketoconazole; betamethasone-17,21-dipropionate; Calcium Dobesilate; Clotrimazole; dexamethasone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Candicort®/ Nizoral® (Experimental): Candicort® is a cream composed by ketoconazole 20mg/g and betamethasone dipropionate 0,64 mg/g that will be dispensed to 80 participants of this group in the first stage. The cream will be applied in the affected area twice a day for 14 (+1) days. In the second stage Nizoral ® will be dispensed to the same participants. It´s a cream composed by ketoconazole 20mg/g that will be applied in the affected area once a day for 14 days. The total duration of treatment may be 28 (+1) days.
  Interventions: Drug: Candicort®; Drug: Nizoral®
- Baycuten N®/ Canesten® (Experimental): Baycuten N® is a cream composed by clotrimazole 10mg and dexamethasone acetate 0.443 mg/g that will be dispensed to 80 participants of this group in the first stage. he cream will be applied in the affected area twice a day for 14 (+1) days. In the second stage Canesten ® will be dispensed to the same participants. It´s a cream composed by clotrimazole 10mg that will be applied in the affected area once a day for 14 days.The total duration of treatment may be 28 (+1) days.
  Interventions: Drug: Baycuten N®; Drug: Canesten®

INTERVENTIONS:
Drug: Candicort® — Apply on the affected area and around it twice a day
  Other Names: ketoconazole and betamethasone dipropionate
  Arms: Candicort®/ Nizoral®
Drug: Nizoral® — Apply on the affected area and around it twice a day
  Other Names: ketoconazole
  Arms: Candicort®/ Nizoral®
Drug: Baycuten N® — Apply on the affected area and around it twice a day
  Other Names: clotrimazole and dexamethasone acetate
  Arms: Baycuten N®/ Canesten®
Drug: Canesten® — Apply on the affected area and around it twice a day
  Other Names: clotrimazole
  Arms: Baycuten N®/ Canesten®

SUMMARY:
To evaluate the no-inferiority of the ketoconazole20mg/g and betamethasone dipropionate 0.64 mg/g association (Candicort®) cream versus clotrimazole 10mg and dexamethasone acetate 0.443 mg/g association (Baycuten N®) cream, general relief of signs and symptoms (erythema, maceration, peeling, blistering / papules / pustules, itching and burning / stinging) 06 (± 1) days after onset treatment.

DETAILED DESCRIPTION:
Candicort® presents formulation with agents that act both etiological agent of superficial mycosis, with coverage for dermatophytes and more frequent yeast; as inflammation generated by the infectious process or prior to it, in cases of secondary fungal infection in wet or potentially infected eczema fungal dermatitis (atopic dermatitis, seborrhoeic dermatitis, intertrigo, dyshidrosis, contact dermatitis).

The active ingredients ketoconazole and betamethasone act, respectively, on the etiologic agent of the infection and the inflammation generated by the process, and the association of both showed a positive therapeutic response in dermatitis with confirmed secondary infections or potential yeast (analysis carried out in association with sulfate neomycin, aimed to cover bacterial infections together).

160 participants that meet all the inclusion criteria and are not classified in any of the exclusion criteria will be randomly allocated to one of two treatment groups(Candicort® or Baycuten N®) of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and consent to participate in this clinical research, expressed by signing the Informed Consent Form (ICF);
* Participants with moderate or severe clinical diagnosis of superficial mycoses caused by Candida ssp or following fungal /dermatophytosis infections: inflammatory tinea corporis inflammatory (except face), inflammatory tinea cruris and inflammatory tinea pedis, with confirmation through direct mycological examination. In moderate or severe superficial mycosis that present at least moderate erythema and itching signs and slight peeling according to the evaluation by the four-point category scale (0=absent, 1-mild, 2-moderate, 3-severe);

Exclusion Criteria:

* Any observational finding (clinical/ physical evaluation) that is interpreted by the investigator as a risk to the research participant's participation in the clinical trial;
* Known hypersensitivity to the drug components used during the study;
* Use of prohibited drugs and treatment prohibited in the last 90 days;
* Immune impairment, according to investigator assessment;
* Vulvovaginal candidiasis diagnostics, balanopreputial, nail, chronic mucocutaneous or oral;
* Diagnosis of chickenpox, rosacea, herpes simplex or zoster, skin tuberculosis or skin syphilis, systemic fungal infection;
* Participants who, though they have studied diagnosis of fungal infections requiring systemic treatment according to the severity of injury and according to the opinion of the investigator;
* Participants that have skin lesions with clinical signs of bacterial infection;
* Participants who, according to investigator assessment, require systemic antibiotic treatment;
* Participants that are in any treatment , in the opinion of the investigator, may affect the results of the study;
* Participants diagnosed with HIV;
* Participants diagnosed with Diabetes Mellitus;
* Participants with a history of smallpox vaccine reaction;
* Women in gestation period or who are breastfeeding;
* Female participants who are in the reproductive age and do not agree to use acceptable methods of contraception (oral contraceptives, injectable contraceptives, intrauterine device (IUD), hormonal implants, barrier methods, hormonal patch and tubal ligation); except surgically sterile (bilateral oophorectomy or hysterectomy), the menopausal for at least one year and participants who declare to perform sexual practices on a not to reproductive way;
* Participant who participated in clinical in the last twelve months, unless the investigator considers that there may be direct benefit to thereof;
* Participant has some kinship of second degree or bond with employees or employees of Sponsor and Research Center.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Percentage change in the total score of signs and symptoms | 6 (±1) days
  Percentage change in the total score of signs and symptoms (erythema, maceration, peeling, blistering /papules /pustules, itching and burning/ stinging) in 6 (±1) days after onset first stage of treatment in relation to the basal.
  The total score will be established by the sum of individual scores of the signs and symptoms assessed by the four-point categorical scale (0=absent, 1=mild, 2=moderate, 3=severe), ranging from 0 to 18 points.
  The percentage change in the total score of signs and symptoms will be calculated by the following expression:
  VTSS(%) = [(TSS0 -TSS6)/ TSS0]*100
  TSS0: total score of signs and symptoms (erythema, maceration, peeling, blistering /papules /pustules, itching and burning/ stinging) in 0 day.
  TSS6: total score of signs and symptoms (erythema, maceration, peeling, blistering /papules /pustules, itching and burning/ stinging) in 6 (±1) days after onset first stage of treatment

SECONDARY OUTCOMES:
Percentage change in the total score of signs and symptoms | 6 (±1) and 14 (+1) days
  Evaluate the percentage change in the total score of signs and symptoms (erythema, maceration, peeling, blistering /papules /pustules, itching and burning/ stinging) during the treatment, evaluated in 6 (±1) and 14 (+1) days after onset first stage of treatment in relation to the basal with the treatment group allocated (Candicort® or Baycuten N®). The total score will be established by the sum of individual scores of the signs and symptoms assessed by the four-point categorical scale (0=absent, 1=mild, 2=moderate, 3=severe), ranging from 0 to 18 points.
Percentage change in the total score of signs and symptoms | Up to 1 month
  Evaluate the percentage change in the total score of signs and symptoms (erythema, maceration, peeling, blistering /papules /pustules, itching and burning/ stinging) in 14 (+1) days after end of the treatment with antifungal isolated (Ketoconazole or Canesten®) in the second stage of treatment. The total score will be established by the sum of individual scores of the signs and symptoms assessed by the four-point categorical scale (0=absent, 1=mild, 2=moderate, 3=severe), ranging from 0 to 18 points.
Mycological cure (Negative result for the direct mycological examination) | Up to 1 month
  Assess the proportion of participants who have mycological cure after completion of treatment with antifungal isolated (Ketoconazole or Canesten®) in 14 (+1) days after end of the treatment with antifungal isolated (Ketoconazole or Canesten®) in the second stage of treatment.
Participants satisfaction regarding the treatment | 6 (±1) days and14 (+1) days
  Assess the satisfaction of participants regarding the treatment using a Visual Analogue Scale (EVA 0 to 100mm) in 6 (±1) and 14 (+1) days after onset first stage of treatment in relation to the basal with the treatment group allocated (Candicort® or Baycuten N®).
Participants satisfaction regarding the treatment | Up to 1 month
  Assess the satisfaction of participants regarding the treatment using a Visual Analogue Scale (EVA 0 to 100mm) in 14 (+1) days after end of the treatment with antifungal isolated (Ketoconazole or Canesten®) in the second stage of treatment.

OTHER OUTCOMES:
Incidence of adverse events | 0 day up to 1 month
  Number of participants with adverse events since first dose of treatment (Candicort® or Baycuten N®) until 30 (+7) days after the end of the second phase of treatment with antifungal isolated (Nizoral® or Canesten®)
Variation in vital signs (heart rate) | 6 (±1) days, 14 (+1) days and up to 1 month
  Variation in heart rate (beats per minute) on each visit from baseline. In this study the physiological parameter for heart rate is 50-100 bpm.
Variation in vital signs (blood pressure) | 6 (±1) days, 14 (+1) days and up to 1 month
  Variation in blood pressure (mmHg) on each visit from baseline. In this study the physiological parameters for systolic blood pressure is ≥ 139 mmHg and diastolic blood pressure is ≤ 89 mmHg.
Rate of participants with any significant variation in Body Mass Index (BMI) | 6 (±1) days, 14 (+1) days and up to 1 month
  Rate of participants with any significant variation in BMI (kg/m2) on each visit, according to investigator assessment.
Rate of participants with any significant variation in physical exam | 6 (±1) days, 14 (+1) days and up to 1 month
  Rate of participants with any significant variation in inspect skin, oropharyngeal system, skeletal muscle system, respiratory system, cardiovascular system, digestive system, genitourinary system, neurological system on each visit, according to investigator assessment.
Rate of participants with any significant variation in complete blood count | Up to 1 month
  Rate of participants with any significant variation in complete blood count on final visit from baseline, according to investigator assessment.
Rate of participants with any significant variation in serum sodium and potassium levels | Up to 1 month
  Rate of participants with any significant variation in serum sodium and potassium (mmol/ L) on final visit from baseline, according to investigator assessment.
Rate of participants with any significant variation in alkaline phosphatase, glutamic oxaloacetic and glutamic pyruvic transaminases levels | Up to 1 month
  Rate of participants with any significant variation in alkaline phosphatase, glutamic oxaloacetic and glutamic pyruvic transaminases (U/L) on final visit from baseline, according to investigator assessment
Rate of participants with any significant variation in bilirubin and fractions levels | Up to 1 month
  Rate of participants with any significant variation in bilirubin and fractions levels (mg/dL) on final visit from baseline, according to investigator assessment.
Rate of participants with any significant variation in serum creatinine and urea levels | Up to 1 month
  Rate of participants with any significant variation in serum creatinine and urea (mg/dL) on final visit from baseline, according to investigator assessment.
Rate of participants with any significant variation in total proteins and fractions levels | Up to 1 month
  Rate of participants with any significant variation in total proteins and fractions (g/dL) on final visit from baseline, according to investigator assessment.
Rate of participants with any significant variation in fasting glycemia level | Up to 1 month
  Rate of participants with any significant variation in fasting glycemia level (mg/dL) on final visit from baseline, according to investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: André Vergnanini, Principal Investigator — Allergisa Pesquisa Dermato-Cosmetica LTDA
Locations (9):
- Brazil (9):
  - Centro de Pesquisa Clínica - CPEC / Associação Obras Sociais Irmã Dulce, Salvador, Estado de Bahia
  - Centro de Pesquisa Clínica do IMIP, Recife, Pernambuco
  - Allergisa Pesquisa Dermato Cosmética Ltda., Campinas, São Paulo
  - Scentryphar Pesquisa Clínica, Campinas, São Paulo
  - Sociedade Campineira de Educação e Instrução - Centro de Pesquisa Clínica São Lucas - PUCCAMP, Campinas, São Paulo
  - Centro de Estudos Multidisciplinar CEPES da Faculdade de Medicina do ABC, Santo André, São Paulo
  - Centro Integrado de Pesquisa - CIP, São José do Rio Preto, São Paulo
  - CDEC Brasil - Centro de Desenvolvimento em Estudo Clínicos Brasil / AFIP-Associação Fundo de Incentivo à pesquisa), São Paulo
  - Centro de Pesquisa Clínica - HSM (Hospital Santa Marcelina), São Paulo